CLINICAL TRIAL: NCT01500733
Title: A Phase II Study of PCI-32765 for Patients With Chronic Lymphocytic Leukemia (CLL) or Small Lymphocytic Lymphoma (SLL) Who Need Therapy and Are Older Than 65 or Have a 17p Deletion
Brief Title: PCI-32765 for Special Cases of Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120035; 12-H-0035
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Leukemia; Leukemia, Lymphocytyc; CLL (Chronic Lymphocytic Leukemia); SLL (Small Lymphocytic Lymphoma)
Keywords: Treatment; CLL (Chronic Lymphocytic Leukemia); SLL (Small Lymphocytic Lymphoma); Leukemia; Lymphocytic Leukemia; Chronic Lymphocytic Leukemia; CLL; Small Lymphocytic Leukemia; SLL
MeSH Terms: conditions — Leukemia; Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Lymphoid | interventions — ibrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elderly greater than 65 (Experimental)
  Interventions: Drug: PCI 32765
- 17p Deletioin (Experimental)
  Interventions: Drug: PCI 32765

INTERVENTIONS:
Drug: PCI 32765 — 420 mg daily

SUMMARY:
Background:

- Chronic lymphocytic leukemia and small lymphocytic lymphoma (CLL/SLL) are types of blood or lymph node cancers that mostly affect the elderly. CLL/SLL both create abnormal white blood cells that hurt the immune system and make it more difficult to fight infections. These cancers are usually diagnosed after age 50; more than half of the people with CLL/SLL are over age 70. Elderly people often do not respond well to standard chemotherapy for CLL/SLL. They may have other health problems that make chemotherapy difficult. In addition, individuals who have a genetic abnormality called 17p deletion also do not respond well to standard treatments for CLL/SLL. Researchers want to test a new cancer treatment drug, PCI-32765, to see if it can treat CLL/SLL in these hard-to-treat groups.

Objectives:

- To see if PCI-32765 is a safe and effective treatment for CLL/SLL in older people and people with 17p deletion.

Eligibility:

* Individuals over 65 years of age who have CLL/SLL.
* Individuals at least 18 years of age who have CLL/SLL and 17p deletion.

Design:

* Participants will be screened with a medical history, physical exam, and imaging studies. Blood and urine samples will be taken. Optional bone marrow and lymph node biopsies may also be taken.
* Participants will take PCI-32765 capsules every day for 28 days (one cycle of treatment). Treatment will be monitored with frequent blood tests and clinic visits.
* PCI-32765 will be given for six cycles of treatment. Those who benefit from the drug will continue to take it as long as there are no side effects and the disease does not progress. Those who do not benefit will stop treatment and have regular followup exams.

DETAILED DESCRIPTION:
CLL/SLL is a malignancy of B cells that predominantly affects the elderly population. Diagnosis is typically made in adults over the age of 50 and more than half of the people with CLL/SLL are over the age of 70. Elderly patients in particular have other comorbidities that limit the tolerability of standard CLL/SLL chemoimmunotherapy regimens and they often have inferior response to these particular regimens. In addition, those patients with a 17p deletion also have inferior outcomes due to rapid progression of disease as well as refractoriness to standard treatment regimens.

It is still unclear what leads to the development of CLL/SLL. However, recent studies indicated that B cell receptor (BCR) signaling is an important contributor to the disease and could be a target for therapy. Bruton s Tyrosine Kinase (Btk) is an enzyme required for BCR signaling.

Ibrutinib is a potent and selective inhibitor of Bruton Tyrosine Kinase (Btk). In vitro lymphoma models have demonstrated that ibrutinib inhibits Btk. Inhibition of Btk blocks downstream BCR signaling pathways and thus prevents B cell proliferation. A phase 1 study of ibrutinib shows activity in multiple lymphomas including CLL/SLL.

This study will investigate the efficacy of ibrutinib for patients with CLL/SLL in patients that are older than 65 who are in need of therapy.This protocol is intended both for patients who have been untreated and those who have undergone other therapies.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Cohort 1: Treated and untreated patients age 65 or older and need for therapy

   Cohort 2: Treated (maximum accrual n=16) and untreated (n=27, evaluable) patients at least 18 years old with 17p deletion or p53 expression by immunohistochemistry or p53 mutation by sequencing analysis.
2. Men and women with histologically confirmed disease as defined by the following:

   * B-lymphocytosis greater than 5000 cells/microL (may be less than 5000 cells/microL if lymphadenopathy is present with histologic confirmation of lymph node involvement by SLL)
   * Immunophenotypic profile read by an expert pathologist as consistent with CLL. This will include CD5, CD19, and CD20 expression by the CLL cells typically also with CD23 expression, but CD23 negative cases may be included if there is no t11;14 translocation present.
3. Active disease as defined by at least one of the following:

   * Weight loss greater than or equal to 10% within the previous 6 months
   * Extreme fatigue
   * Fevers of greater than 100.5 degrees F for greater than or equal to 2 weeks without evidence of infection
   * Night sweats for more than one month without evidence of infection
   * Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia and/or thrombocytopenia
   * Massive or progressive splenomegaly
   * Massive nodes or clusters or progressive lymphadenopathy
   * Progressive lymphocytosis with an increase of greater than 50% over a 2 month period, or an anticipated doubling time of less than 6 months
   * Compensated autoimmune hemolysis
4. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2
5. ANC greater than 500/microL, platelets greater than 30,000/microL
6. Agreement to use contraception during the study and for 90 days after the last dose of study drug if sexually active and able to bear children
7. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty
8. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local subject privacy regulations)

EXCLUSION CRITERIA:

1. Previous radiotherapy, radioimmunotherapy, biological therapy, chemotherapy, or treatment with an investigational product fpr CCL treatement in the last 4 weeks (i.e. intravenous immunoglobulin).
2. Transformed CLL
3. Autoimmune hemolytic anemia or thrombocytopenia requiring steroid therapy
4. Impaired hepatic function: Total bilirubin greater than or equal to 1.5 times upper limit of normal unless dute to Gilbert's disease, AST/ ALT greater than or equal to 2.5 times institutional upper limit of normal unless due to infiltration of the liver.
5. Impaired renal funtion: Creatinine greater than or equal to 2.0 mg/dL or GFR less than or equal to 50ml/min
6. Life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the subject's safety, interfere with the absorption or metabolism of PCI-32765 PO, or put the study outcomes at undue risk
7. Concomitant immunotherapy, chemotherapy, radiotherapy, corticosteroids (at dosages equivalent to prednisone > 20 mg/day), or experimental therapy
8. Active Hepatitis B infection
9. HIV infection
10. Female patients: Current pregnancy or unwilling to take oral contraceptives or refrain from pregnancy if of childbearing potential or currently breastfeeding. Male patients who are unwilling to follow the contraception requirements described in this protocol.
11. Psychiatric illness/social situations that would limit the patient s ability to tolerate and/or comply with study requirements.
12. Unable to understand the investigational nature of the study or give informed consent.
13. Individuals < 18 yrs old
14. Known hypersensitivity to any component of PCI-32765
15. Any prior therapy with PCI 32765 or any other BTK inhibitors.
16. Requires anticoagulation with warfarin.
17. Requires treatment with strong CY3A4/5 and/or CYP2D6 inhibitors (unless no alternative is available).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2012-01-05 (Actual); Primary Completion 2014-06-20 (Actual); Study Completion 2034-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Andy Itsara, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Harris NL, Jaffe ES, Diebold J, Flandrin G, Muller-Hermelink HK, Vardiman J. Lymphoma classification--from controversy to consensus: the R.E.A.L. and WHO Classification of lymphoid neoplasms. Ann Oncol. 2000;11 Suppl 1:3-10. PMID 10707771
- [Background] Hallek M, Cheson BD, Catovsky D, Caligaris-Cappio F, Dighiero G, Dohner H, Hillmen P, Keating MJ, Montserrat E, Rai KR, Kipps TJ; International Workshop on Chronic Lymphocytic Leukemia. Guidelines for the diagnosis and treatment of chronic lymphocytic leukemia: a report from the International Workshop on Chronic Lymphocytic Leukemia updating the National Cancer Institute-Working Group 1996 guidelines. Blood. 2008 Jun 15;111(12):5446-56. doi: 10.1182/blood-2007-06-093906. Epub 2008 Jan 23. PMID 18216293
- [Background] Rawstron AC, Bennett FL, O'Connor SJ, Kwok M, Fenton JA, Plummer M, de Tute R, Owen RG, Richards SJ, Jack AS, Hillmen P. Monoclonal B-cell lymphocytosis and chronic lymphocytic leukemia. N Engl J Med. 2008 Aug 7;359(6):575-83. doi: 10.1056/NEJMoa075290. PMID 18687638
- [Result] Ahn IE, Farooqui MZH, Tian X, Valdez J, Sun C, Soto S, Lotter J, Housel S, Stetler-Stevenson M, Yuan CM, Maric I, Calvo KR, Nierman P, Hughes TE, Saba NS, Marti GE, Pittaluga S, Herman SEM, Niemann CU, Pedersen LB, Geisler CH, Childs R, Aue G, Wiestner A. Depth and durability of response to ibrutinib in CLL: 5-year follow-up of a phase 2 study. Blood. 2018 May 24;131(21):2357-2366. doi: 10.1182/blood-2017-12-820910. Epub 2018 Feb 26. PMID 29483101
- [Derived] Itsara A, Rogness VM, Samples L, Yuan CM, Wang HW, Ahn IE, Farooqui MZH, Tian X, Sun C, Tomasulo E, Soto S, Superata J, Bezkorovaynaya L, Hughes TE, Nierman PK, Wiestner A. A Decade of Ibrutinib for CLL with and without TP53 Aberration: Final Report on an Investigator-Sponsored Phase 2 Study. Blood. 2025 Dec 17:blood.2025029971. doi: 10.1182/blood.2025029971. Online ahead of print. PMID 41405491
- [Derived] Alsadhan A, Chen J, Gaglione EM, Underbayev C, Tuma PL, Tian X, Freeman LA, Baskar S, Nierman P, Soto S, Itsara A, Ahn IE, Sun C, Bibikova E, Hartmann TN, Mhibik M, Wiestner A. CD49d Expression Identifies a Biologically Distinct Subtype of Chronic Lymphocytic Leukemia with Inferior Progression-Free Survival on BTK Inhibitor Therapy. Clin Cancer Res. 2023 Sep 15;29(18):3612-3621. doi: 10.1158/1078-0432.CCR-22-3217. PMID 37227160
- [Derived] Cyr MG, Mhibik M, Qi J, Peng H, Chang J, Gaglione EM, Eik D, Herrick J, Venables T, Novick SJ, Courouble VV, Griffin PR, Wiestner A, Rader C. Patient-derived Siglec-6-targeting antibodies engineered for T-cell recruitment have potential therapeutic utility in chronic lymphocytic leukemia. J Immunother Cancer. 2022 Nov;10(11):e004850. doi: 10.1136/jitc-2022-004850. PMID 36442911
- [Derived] Allan JN, Shanafelt T, Wiestner A, Moreno C, O'Brien SM, Li J, Krigsfeld G, Dean JP, Ahn IE. Long-term efficacy of first-line ibrutinib treatment for chronic lymphocytic leukaemia in patients with TP53 aberrations: a pooled analysis from four clinical trials. Br J Haematol. 2022 Feb;196(4):947-953. doi: 10.1111/bjh.17984. Epub 2021 Dec 5. PMID 34865212
- [Derived] Brieghel C, Aarup K, Torp MH, Andersen MA, Yde CW, Tian X, Wiestner A, Ahn IE, Niemann CU. Clinical Outcomes in Patients with Multi-Hit TP53 Chronic Lymphocytic Leukemia Treated with Ibrutinib. Clin Cancer Res. 2021 Aug 15;27(16):4531-4538. doi: 10.1158/1078-0432.CCR-20-4890. Epub 2021 May 7. PMID 33963002
- [Derived] Ahn IE, Underbayev C, Albitar A, Herman SE, Tian X, Maric I, Arthur DC, Wake L, Pittaluga S, Yuan CM, Stetler-Stevenson M, Soto S, Valdez J, Nierman P, Lotter J, Xi L, Raffeld M, Farooqui M, Albitar M, Wiestner A. Clonal evolution leading to ibrutinib resistance in chronic lymphocytic leukemia. Blood. 2017 Mar 16;129(11):1469-1479. doi: 10.1182/blood-2016-06-719294. Epub 2017 Jan 3. PMID 28049639
- [Derived] Ahn IE, Jerussi T, Farooqui M, Tian X, Wiestner A, Gea-Banacloche J. Atypical Pneumocystis jirovecii pneumonia in previously untreated patients with CLL on single-agent ibrutinib. Blood. 2016 Oct 13;128(15):1940-1943. doi: 10.1182/blood-2016-06-722991. Epub 2016 Aug 8. PMID 27503501
- [Derived] Bitar C, Farooqui MZ, Valdez J, Saba NS, Soto S, Bray A, Marti G, Wiestner A, Cowen EW. Hair and Nail Changes During Long-term Therapy With Ibrutinib for Chronic Lymphocytic Leukemia. JAMA Dermatol. 2016 Jun 1;152(6):698-701. doi: 10.1001/jamadermatol.2016.0225. PMID 26982511
- [Derived] Lipsky AH, Farooqui MZ, Tian X, Martyr S, Cullinane AM, Nghiem K, Sun C, Valdez J, Niemann CU, Herman SE, Saba N, Soto S, Marti G, Uzel G, Holland SM, Lozier JN, Wiestner A. Incidence and risk factors of bleeding-related adverse events in patients with chronic lymphocytic leukemia treated with ibrutinib. Haematologica. 2015 Dec;100(12):1571-8. doi: 10.3324/haematol.2015.126672. Epub 2015 Oct 1. PMID 26430171
- [Derived] Sun C, Tian X, Lee YS, Gunti S, Lipsky A, Herman SE, Salem D, Stetler-Stevenson M, Yuan C, Kardava L, Moir S, Maric I, Valdez J, Soto S, Marti GE, Farooqui MZ, Notkins AL, Wiestner A, Aue G. Partial reconstitution of humoral immunity and fewer infections in patients with chronic lymphocytic leukemia treated with ibrutinib. Blood. 2015 Nov 5;126(19):2213-9. doi: 10.1182/blood-2015-04-639203. Epub 2015 Sep 3. PMID 26337493
- [Derived] Farooqui MZ, Valdez J, Martyr S, Aue G, Saba N, Niemann CU, Herman SE, Tian X, Marti G, Soto S, Hughes TE, Jones J, Lipsky A, Pittaluga S, Stetler-Stevenson M, Yuan C, Lee YS, Pedersen LB, Geisler CH, Calvo KR, Arthur DC, Maric I, Childs R, Young NS, Wiestner A. Ibrutinib for previously untreated and relapsed or refractory chronic lymphocytic leukaemia with TP53 aberrations: a phase 2, single-arm trial. Lancet Oncol. 2015 Feb;16(2):169-76. doi: 10.1016/S1470-2045(14)71182-9. Epub 2014 Dec 31. PMID 25555420
- [Derived] Herman SE, Niemann CU, Farooqui M, Jones J, Mustafa RZ, Lipsky A, Saba N, Martyr S, Soto S, Valdez J, Gyamfi JA, Maric I, Calvo KR, Pedersen LB, Geisler CH, Liu D, Marti GE, Aue G, Wiestner A. Ibrutinib-induced lymphocytosis in patients with chronic lymphocytic leukemia: correlative analyses from a phase II study. Leukemia. 2014 Nov;28(11):2188-96. doi: 10.1038/leu.2014.122. Epub 2014 Apr 4. PMID 24699307
- [Derived] Herman SE, Mustafa RZ, Gyamfi JA, Pittaluga S, Chang S, Chang B, Farooqui M, Wiestner A. Ibrutinib inhibits BCR and NF-kappaB signaling and reduces tumor proliferation in tissue-resident cells of patients with CLL. Blood. 2014 May 22;123(21):3286-95. doi: 10.1182/blood-2014-02-548610. Epub 2014 Mar 21. PMID 24659631
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-H-0035.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Elderly Cohort: Chronic lymphocytic leukemia patients 65 years or older
- TP53 Cohort: Chronic lymphocytic leukemia patients having TP53 aberration, either due to deletion of chromosome 17p or TP53 mutation
Period: Overall Study
Arm/Group | Elderly Cohort | TP53 Cohort
Started | 35 | 51
Completed | 33 | 48
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly Cohort | TP53 Cohort | Total
Number analyzed (Participants) | 35 | 51 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 30 | 31
  >=65 years | 34 | 21 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 20 | 36
  Male | 19 | 31 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 35 | 48 | 83
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 33 | 44 | 77
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate at 6 Months
Description: The primary endpoint was response after 6 cycles of therapy. Overall response rate was calculated as complete response plus partial response, based on the International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2008 criteria.as follows:
  Complete response (CR): all group A and group B criteria are met
  * Group A criteria: resolution of enlarged lymph nodes, normal size spleen and liver, absolute lymphocyte count < 4,000/uL, normocellular bone marrow with < 30% lymphocytes without nodules
  * Group B criteria: improved blood count (platelet count > 100,000/uL, hemoglobin > 11.0 g/dL, neutrophils > 1,500/uL)
  Partial response (PR): at least 2 of the group A criteria plus one of the group B criteria are met
  * Group A criteria: >=50% decrease in target lymph nodes, >=50% decrease in spleen size, >=50% decrease in liver size, 50% reduction in marrow infiltrates
  * Group B criteria: platelet count > 100,000/uL, hemoglobin > 11.0 g/dL, neutrophils > 1,500/uL
Time Frame: 6 months
Population: The analyses included only those subjects who received ibrutinib, and completed 6 cycles of therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Elderly Cohort | TP53 Cohort
Number analyzed (Participants) | 33 | 48
percentage of participants | 93.9 [79.8 to 99.3] | 95.8 [85.7 to 99.5]

ADVERSE EVENTS:
Time Frame: 69 months
Groups:
- TP53 Cohort: Chronic lymphocytic leukemia patients having T53 aberration, either due to deletion of chromosome 17p or TP53 mutation
Arm/Group | Elderly Cohort | TP53 Cohort
All-Cause Mortality (participants affected / at risk) | 5/35 | 13/51
Serious Adverse Events (participants affected / at risk) | 25/35 | 29/51
Other Adverse Events (participants affected / at risk) | 35/35 | 51/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elderly Cohort (N=35) | TP53 Cohort (N=51)
Anemia (Blood and lymphatic system disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 4
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 3
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Heart failure (Cardiac disorders) | 1 | 1
Stroke (Cardiac disorders) | 0 | 1
Retinopathy (Eye disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Death, NOS (General disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 0
Fever (General disorders) | 0 | 2
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0
Immune system disorders - Other, specify (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 5 | 7
Lung infection (Infections and infestations) | 9 | 7
Pleural infection (Infections and infestations) | 0 | 1
Prostate infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 3
Skin infection (Infections and infestations) | 1 | 3
Upper respiratory infection (Infections and infestations) | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 9
Amnesia (Nervous system disorders) | 0 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Elderly Cohort (N=35) | TP53 Cohort (N=51)
Anemia (Blood and lymphatic system disorders) | 29 | 40
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 | 8
Leukocytosis (Blood and lymphatic system disorders) | 12 | 20
Lymph node pain (Blood and lymphatic system disorders) | 2 | 8
Atrial fibrillation (Cardiac disorders) | 7 | 8
Atrioventricular block first degree (Cardiac disorders) | 0 | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 3
Chest pain - cardiac (Cardiac disorders) | 1 | 0
Hypertension (Cardiac disorders) | 2 | 0
Palpitations (Cardiac disorders) | 7 | 10
Pericardial effusion (Cardiac disorders) | 2 | 0
Sinus bradycardia (Cardiac disorders) | 6 | 9
Sinus tachycardia (Cardiac disorders) | 2 | 6
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 5 | 2
Ear pain (Ear and labyrinth disorders) | 1 | 2
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 4 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 3 | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 | 3
Hypothyroidism (Endocrine disorders) | 1 | 0
Blurred vision (Eye disorders) | 3 | 4
Cataract (Eye disorders) | 5 | 1
Conjunctivitis (Eye disorders) | 1 | 5
Dry eye (Eye disorders) | 2 | 5
Eye disorders - Other, specify (Eye disorders) | 9 | 14
Eye pain (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 2 | 1
Glaucoma (Eye disorders) | 1 | 1
Scleral disorder (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 2
Watering eyes (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 7
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anorexia (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 2 | 4
Cheilitis (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 6 | 3
Dental caries (Gastrointestinal disorders) | 1 | 3
Diarrhea (Gastrointestinal disorders) | 25 | 35
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 4
Flatulence (Gastrointestinal disorders) | 2 | 2
Gastritis (Gastrointestinal disorders) | 1 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 7 | 7
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 11 | 13
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 6 | 12
Nausea (Gastrointestinal disorders) | 6 | 12
Oral hemorrhage (Gastrointestinal disorders) | 3 | 2
Oral pain (Gastrointestinal disorders) | 0 | 1
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 3 | 8
Chills (General disorders) | 8 | 12
Dizziness (General disorders) | 0 | 2
Edema face (General disorders) | 1 | 1
Edema limbs (General disorders) | 11 | 18
Fatigue (General disorders) | 12 | 23
Fever (General disorders) | 7 | 16
Flu like symptoms (General disorders) | 3 | 7
General disorders and administration site conditions - Other, specify (General disorders) | 5 | 7
Headache (General disorders) | 0 | 1
Infusion site extravasation (General disorders) | 0 | 1
Localized edema (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 2
Neck edema (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 3 | 4
Pain (General disorders) | 15 | 19
Weight loss (General disorders) | 1 | 0
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 2 | 0
Allergic reaction (Immune system disorders) | 1 | 5
Anorectal infection (Infections and infestations) | 0 | 1
Bronchial infection (Infections and infestations) | 4 | 7
Eye infection (Infections and infestations) | 1 | 2
Gum infection (Infections and infestations) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 14 | 29
Laryngitis (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 8 | 5
Nail infection (Infections and infestations) | 2 | 3
Otitis externa (Infections and infestations) | 2 | 0
Papulopustular rash (Infections and infestations) | 6 | 4
Paronychia (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 0 | 1
Rhinitis infective (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 14 | 14
Skin infection (Infections and infestations) | 9 | 10
Upper respiratory infection (Infections and infestations) | 17 | 18
Urinary tract infection (Infections and infestations) | 5 | 7
Vaginal infection (Infections and infestations) | 1 | 0
Vulval infection (Infections and infestations) | 1 | 1
Bruising (Injury, poisoning and procedural complications) | 25 | 34
Fall (Injury, poisoning and procedural complications) | 7 | 9
Fracture (Injury, poisoning and procedural complications) | 4 | 2
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 4 | 8
Intraoperative skin injury (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 4 | 5
Alanine aminotransferase increased (Investigations) | 12 | 22
Alkaline phosphatase increased (Investigations) | 10 | 12
Aspartate aminotransferase increased (Investigations) | 13 | 15
Blood bilirubin increased (Investigations) | 9 | 18
Cardiac troponin I increased (Investigations) | 0 | 1
CPK increased (Investigations) | 5 | 6
Creatinine increased (Investigations) | 17 | 28
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 | 3
Haptoglobin decreased (Investigations) | 3 | 4
Hypercalcemia (Investigations) | 1 | 0
Hypermagnesemia (Investigations) | 0 | 1
Hypernatremia (Investigations) | 0 | 1
Hypoalbuminemia (Investigations) | 0 | 1
Hyponatremia (Investigations) | 1 | 0
INR increased (Investigations) | 4 | 2
Investigations - Other, specify (Investigations) | 8 | 5
Lipase increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 15 | 19
Lymphocyte count increased (Investigations) | 32 | 48
Neutrophil count decreased (Investigations) | 20 | 34
Platelet count decreased (Investigations) | 28 | 38
Weight gain (Investigations) | 17 | 28
Weight loss (Investigations) | 7 | 11
White blood cell decreased (Investigations) | 11 | 11
Alkalosis (Metabolism and nutrition disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 10 | 8
Dehydration (Metabolism and nutrition disorders) | 2 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 5 | 10
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 5 | 7
Hypernatremia (Metabolism and nutrition disorders) | 15 | 17
Hyperuricemia (Metabolism and nutrition disorders) | 15 | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 | 26
Hypocalcemia (Metabolism and nutrition disorders) | 17 | 23
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 6 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 6
Hyponatremia (Metabolism and nutrition disorders) | 8 | 10
Hypophosphatemia (Metabolism and nutrition disorders) | 9 | 13
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 | 2
Obesity (Metabolism and nutrition disorders) | 5 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 23
Arthritis (Musculoskeletal and connective tissue disorders) | 11 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 4 | 10
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 19
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 4
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 20
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 | 8
Amnesia (Nervous system disorders) | 1 | 1
Dizziness (Nervous system disorders) | 3 | 16
Dysarthria (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 6 | 10
Lethargy (Nervous system disorders) | 0 | 1
Memory impairment (Nervous system disorders) | 1 | 3
Nervous system disorders - Other, specify (Nervous system disorders) | 2 | 3
Neuralgia (Nervous system disorders) | 1 | 1
Paresthesia (Nervous system disorders) | 4 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 3
Presyncope (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Sinus pain (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Transient ischemic attacks (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 1
Vasovagal reaction (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 3
Confusion (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 4 | 3
Psychiatric disorders - Other, specify (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Hematuria (Renal and urinary disorders) | 6 | 10
Hemoglobinuria (Renal and urinary disorders) | 1 | 4
Proteinuria (Renal and urinary disorders) | 2 | 2
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 4 | 5
Renal colic (Renal and urinary disorders) | 1 | 0
Urinary frequency (Renal and urinary disorders) | 2 | 3
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Urine discoloration (Renal and urinary disorders) | 0 | 1
Ejaculation disorder (Reproductive system and breast disorders) | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0
Perineal pain (Reproductive system and breast disorders) | 0 | 1
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 2 | 1
Vaginal pain (Reproductive system and breast disorders) | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 15 | 19
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 10
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 10
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 2
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 4
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 5
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 | 3
Nail loss (Skin and subcutaneous tissue disorders) | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 2 | 6
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 5
Purpura (Skin and subcutaneous tissue disorders) | 5 | 4
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 25
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 27 | 40
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 4
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 5 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 11 | 2
Hematoma (Vascular disorders) | 3 | 2
Hot flashes (Vascular disorders) | 1 | 7
Hypertension (Vascular disorders) | 12 | 23
Hypotension (Vascular disorders) | 1 | 2
Lymphedema (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 2
Thromboembolic event (Vascular disorders) | 0 | 1
Vascular disorders - Other, specify (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes